CLINICAL TRIAL: NCT05842382
Title: Effect of High Dose Intravenous Vitamin C as an Adjunct in the Treatment of Patients With Severe Pneumonia in Intensive Care Unit: a Multi-center, Double-blinded, Two-arm, Placebo-controlled, Randomized Trial
Brief Title: Effect of High Dose Intravenous Vitamin C in Severe Pneumonia
Acronym: VICSEP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Ain Medicare Sdn Bhd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VICSEP
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Pneumonia
Keywords: Severe pneumonia; Critically ill; Ascorbic acid; Vitamin C; Mechanical ventilation; Ventilation-free day
MeSH Terms: conditions — Pneumonia; Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV Vitamin C (12g/day) (Experimental): IV Vitamin C 3g diluted with dextrose 5% into 50ml, given every 6 hourly (12g/day), infused over 30 minutes under close monitoring, until successful extubation (minimum 16 doses, maximum 40 doses).
  Interventions: Drug: Active Ingredient
- Placebo (Placebo Comparator): IV dextrose 5% 50ml, given every 6 hourly, infused over 30 minutes under close monitoring, until successful extubation (minimum 16 doses, maximum 40 doses).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active Ingredient — IV Vitamin C (12g/day)
  Arms: IV Vitamin C (12g/day)
Drug: Placebo — IV dextrose 5%
  Arms: Placebo

SUMMARY:
This trial is a multicenter, randomized, double-blind, two-arm, parallel-group, placebo-controlled trial to investigate the effect of high dose intravenous (IV) Vitamin C as an adjunct to the standard of care for patients with severe pneumonia versus placebo in ICU.

DETAILED DESCRIPTION:
Subjects will be randomized 1:1 to receive either high dose IV Vitamin C (12g/day) or placebo, every 6 hourly, until successful extubation (minimum 16 doses, maximum 40 doses). Placebo will be the equivalent volume of dextrose 5% given intravenously. Active drug or placebo will be prepared in a sterile method by designated personnel at each site. Active drug or placebo will be prepared in a 50cc syringe and infusion tubing attached, where both are coloured and UV-protected. The recruitment period is expected to be 24 months. Phone call follow-up will be conducted at day 60 (+7 days) post-randomization to review subjects' activities of daily living. All data will be entered electronically into REDCap.

All randomized subjects will be included in the intention-to-treat analysis (ITT) dataset for primary and secondary efficacy endpoints analyses. Safety analysis will be conducted for all subjects who received at least one dose of study drug. There are no interim analyses planned in this trial. At least one safety review will be conducted at 50% target recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are aged 18 and above
* Patients who are diagnosed with severe pneumonia
* Patients who are mechanically ventilated

Exclusion Criteria:

* Known allergy to Vitamin C
* Pregnancy
* Known history of ongoing concomitant infection
* Participation in another clinical trial and/or receipt of investigational drugs within 4 weeks prior to enrollment
* Moribund patient with multiorgan failure to the judgement of the treating physician, who is not expected to survive 24 hours
* Patient who requires home oxygen therapy or mechanical ventilation, including tracheostomy or non-invasive ventilation, except for CPAP/BIPAP for sleep-disordered breathing
* Known history of previous or current diagnosis of renal stones
* Known diagnosis of glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Known diagnosis of hemochromatosis
* Known diagnosis of poorly controlled chronic pulmonary disease, including:

  * Chronic obstructive pulmonary disease with oxygen therapy
  * Chronic restrictive pulmonary disease with oxygen therapy
  * Bronchial asthma on Step 5 of treatment ladder as shown in Pocket Guide for Asthma Management and Prevention
  * Lung cancer in Stage IV of disease
* Known diagnosis of heart failure on anti-failure treatment or requiring mechanical hemodynamic support (e.g. LVAD), with recent hospitalization within 3 months (90 days) from the date of current admission.
* Immunocompromised state
* Known diagnosis of malignancy and ongoing chemotherapy or radiotherapy as there is evidence that antioxidant supplement before and during treatment was associated with an increased hazard of recurrence
* Known diagnosis of malignancy who had completed chemotherapy or radiotherapy with absolute neutrophil count ≤100 cells/mm3
* Known diagnosis of Stage 4 and above chronic kidney disease (GFR <30 ml/min/1.73m2) and end-stage renal disease on regular dialysis (including peritoneal dialysis or hemodialysis)
* Known history of renal transplantation
* Absence of family members or next of kin for informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Ventilation-free days (VFD) at 28-days | First 28 days after start of randomization
  Unit of measurement: Ventilation-free days

SECONDARY OUTCOMES:
Subdistribution hazard ratio of ventilation-free event with mortality as the competing event | First 28 days after start of randomization
  Unit of measurement: Cumulative incidence curve, Subdistribution hazard ratio
Sequential Organ Failure Assessment (SOFA) score | Baseline, Day 4, Post intervention
  Unit of measurement: Point score
Plasma C-reactive protein (CRP) level | Baseline, Day 4, Post intervention
  Unit of measurement: mg/L
28-day vasopressor-free days | First 28 days after start of randomization
  Unit of measurement: Vasopressor-free day
28-day intensive care unit-free days | First 28 days after start of randomization
  Unit of measurement: ICU-free days
60-day hospitalization-free days | First 60 days after start of randomization
  Unit of measurement: Hospitalization-free days
All-cause mortality rates at 28-day | First 28 days after start of randomization
  Unit of measurement: Proportion, Percentage
Barthel index of activities of daily living | Baseline, Day 60
  Unit of measurement: Point score
Plasma ascorbate levels | Baseline, Day 2 (Between 8th and 9th dose OR Between 9th and 10th dose)
  Unit of measurement: μM

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Wong Ke Wen, MBBS MRCP, Principal Investigator — Hospital Umum Sarawak, Malaysia
Locations (3):
- Malaysia (3):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak

IPD SHARING:
Plan to Share IPD: No